CLINICAL TRIAL: NCT05557591
Title: A Phase 2 Study of Cemiplimab (Anti-PD-1 Antibody) in Combination With BNT116 (FixVac Lung) Versus Cemiplimab Monotherapy in First-Line Treatment of Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) With Tumors Expressing PD-L1 ≥50%
Brief Title: A Trial to Learn How the Cancer Vaccine BNT116 in Combination With Cemiplimab Works and How Safe the Combination is in Adults With Advanced Non-small Cell Lung Cancer (EMPOWERVAX Lung 1)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-2045; 2021-006901-31 (EudraCT Number); 2023-503221-19-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Cancer Vaccine; Immunotherapy; Programmed cell death ligand-1 (PD-L1) monoclonal antibody; Treatment naïve Advanced Non-Small Cell Lung Cancer (NSCLC); EMPOWERVAX Lung 1
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 2: Cemiplimab (Experimental): Arm A: Cemiplimab is administered by IV infusion Q3W
  Interventions: Drug: Cemiplimab
- Phase 2: BNT116 + Cemiplimab (Experimental): Arm B: BNT116 is administered by IV injection. Cemiplimab is administered by IV infusion Q3W.
  Interventions: Drug: BNT116; Drug: Cemiplimab

INTERVENTIONS:
Drug: BNT116 — BNT116 is administered by IV injection.
  Arms: Phase 2: BNT116 + Cemiplimab
Drug: Cemiplimab — Cemiplimab is administered Q3W by IV infusion
  Other Names: REGN2810; Libtayo

SUMMARY:
This study is researching an investigational drug, called BNT116, in combination with cemiplimab. BNT116 and cemiplimab will each be called a "study drug", and together be called "study drugs". The study is focused on patients who have advanced non-small cell lung cancer (NSCLC).

The aims of this study are to see how safe and tolerable BNT116 is in combination with cemiplimab and to see how effective BNT116 in combination with cemiplimab is compared to cemiplimab by itself at treating cancer.

The study is looking at several other research questions, including:

* What side effects may happen from receiving the study drugs
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug(s) (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria

1. Participants with non-squamous or squamous histology NSCLC with stage IIIB or stage IIIC disease who are not candidates for surgical resection or definitive chemoradiation per investigator assessment or stage IV (metastatic) disease who received no prior systemic treatment for recurrent or metastatic NSCLC
2. Availability of an archival or on-study obtained formalin-fixed, paraffin-embedded tumor tissue sample as defined in the protocol.
3. Expression of Programmed cell death ligand-1 (PD-L1) ≥50%, as described in the protocol.
4. Participants must have at least 1 radiographically measurable lesion by computerized tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) criteria
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤1

Key Exclusion Criteria

1. Participants who have never smoked, defined as smoking ≤100 cigarettes in a lifetime
2. Active or untreated brain metastases or spinal cord compression. Participants are eligible if central nervous system (CNS) metastases are adequately treated and patients have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment
3. Participants with tumors tested positive for epidermal growth factor receptor (EGFR) gene mutations, anaplastic lymphoma kinase (ALK) gene translocations, or C-ros oncogene receptor tyrosine kinase 1 (ROS1) fusions
4. Encephalitis, meningitis, or uncontrolled seizures in the year prior to enrollment
5. Participants with history of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), of active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or of pneumonitis within the last 5 years
6. Prior splenectomy
7. Uncontrolled infection with human immunodeficiency virus (HIV), HBV or hepatitis C infection (HCV); or diagnosis of immunodeficiency as defined in the protocol
8. Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk of immune-related treatment-emergent adverse events (imTEAEs)
9. Participants requiring corticosteroid therapy (>5 mg prednisone/day or equivalent) within 14 days of randomization
10. Another malignancy that is progressing or requires treatment, except for non melanomatous skin cancer that has undergone potentially curative therapy, in situ cervical carcinoma, or any other localized tumor that has been treated, and the participant is deemed to be in complete remission for at least 2 years prior to enrollment, and no additional therapy is required during the study period
11. Documented or suspected ongoing severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as defined in the protocol
12. Patients who have received prior systemic therapies for NSCLC are excluded except for of the following:

    1. Adjuvant or neoadjuvant platinum-based doublet chemotherapy (after surgery and/or radiation therapy) if recurrent or metastatic disease develops more than 6 months after completing therapy if toxicities have resolved to CTCAE grade ≤1 or baseline except for alopecia and peripheral neuropathy.
    2. Anti-PD-(L)1 with or without LAG-3 as an adjuvant or neoadjuvant therapy as long as the last dose is >12 months prior to enrollment.
    3. Prior exposure to other immunomodulatory or vaccine therapies as an adjuvant or neoadjuvant therapy such as anti-cytotoxic T lymphocyte-associated antigen (anti-CTLA-4) antibodies if the last dose is >6 months prior to enrollment
13. History or current evidence of significant cardiovascular disease including, myocarditis, congestive heart failure (as defined by New York Heart Association Functional Classification III and IV), unstable angina, serious uncontrolled arrhythmia, and myocardial infarction 6 months prior to study enrollment.
14. Hypersensitivity to cemiplimab or BNT116 or any of their excipients, or contraindicated to cemiplimab per approved local labeling.
15. Patients treated with immunostimulatory agents that may influence the efficacy of the investigational medicinal products (IMPs) are not allowed if they received such agents within 6 weeks or five halve lives of the drug.

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2028-01-26 (Estimated); Study Completion 2028-05-16 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as assessed by blinded independent review committee (BIRC) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) | Up to 136 weeks from randomization
  Proportion of patients with a best overall response of confirmed complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
ORR by investigator assessment | Up to 136 weeks from randomization
  Proportion of patients with a best overall response of confirmed CR or PR
Duration of Response (DOR) as assessed by BIRC using RECIST 1.1 | Up to 3 years from last patient randomized
  The time from first response of CR or PR to first radiographic progression or death due to any cause for patients with confirmed CR or PR
DOR by investigator assessment | Up to 3 years from last patient randomized
  The time from first response of CR or PR to first radiographic progression or death due to any cause for patients with confirmed CR or PR
Progression Free Survival (PFS) as assessed by BIRC using RECIST 1.1 | Up to 3 years from last patient randomized
  The time from randomization to the date of the first radiographic progression or death due to any cause, whichever occurred earlier
PFS by investigator assessment | Up to 3 years from last patient randomized
  The time from randomization to the date of the first radiographic progression or death due to any cause, whichever occurred earlier
Overall Survival (OS) | Up to 3 years from last patient randomized
  The time from enrollment to the date of death due to any cause
Incidence of treatment-emergent adverse events (TEAEs) | Up to 3 years
  A TEAE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Incidences of serious adverse events (SAEs) | Up to 3 years
  An SAE is any untoward medical occurrence that at any dose:
  * Results in death - includes all deaths, even those that appear to be completely unrelated to study drug (eg, a car accident in which a patient is a passenger)
  * Is life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event
Incidences of deaths | Up to 3 years
Incidences of laboratory abnormalities | Up to 3 years
  According to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Causality grading system (≥ Grade 3 or higher)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (52):
- United States (9):
  - The Oncology Institute of Hope and Innovation, Los Angeles, California
  - UCLA Medical Center, Santa Monica, California
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - San Juan Oncology Associates, Farmington, New Mexico
  - Weill Cornell Medicine, New York, New York
  - FirstHealth of the Carolinas Outpatient Cancer Center, Pinehurst, North Carolina
  - Millenium Research & Clinical Development, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Georgia (6):
  - LTD High Technology Hospital Medcenter, Batumi
  - LLC Todua Clinic, Tbilisi
  - LTD New Hospitals, Tbilisi
  - LTD Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
  - LTD Cancer Research Centre, Tbilisi
  - Caucasus Medical Centre, Tbilisi
- Germany (5):
  - Staedtisches Klinikum Muenchen Bogenhausen, München, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt, Frankfurt
  - Universitaetsklinikum Giessen Und Marburg Gmbh Standort Giessen, Giessen
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Klinikverbund Kempten-Oberallgäu, Kempten
- South Korea (7):
  - Korea University Anam Hospital, Seoul, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - National Cancer Center Korea, Goyang
  - Asan Medical Center, Seoul
  - Yonsei Severance, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (11):
  - Catalan Institute of Oncology Badalona, Badalona, Barcelona
  - Althaia Xarxa Assistencial Universitaria Manresa, Manresa, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Hospital General Universitario Gregorio Marañon (HGUGM), Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen del Rocio, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (5):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Tzu Chi Hospital, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (9):
  - Adana Medical Park Seyhan Hospital, Adana, Adana
  - Baskent University, Yüreğir, Adana
  - Yeditepe University Kosuyolu Hospital, Kadıköy, Istanbul
  - Ege University Faculty of Medicine, Bornova, İzmir
  - Ozel Liv Hospital, Ankara
  - Sbu Doctor Abdurrahman Yurtaslan Ankara Onkoloji Suam, Ankara
  - Bezmialem Foundation University Medical Faculty, Istanbul
  - Istanbul Medeniyet University - Prof Dr Suleyman Yalcin Sehir Hospital, Istanbul
  - Izmir Economy University Medical Point Hospital, Izmir

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/